CLINICAL TRIAL: NCT02272036
Title: Improvement of Colonoscopy Preparation by New Media (SMS) (PERICLES-II-Study)
Brief Title: Short Message Service in Colonoscopy Preparation (PERICLES-II-SMS)
Acronym: PERICLES-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 102014
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Colon Cancer
Keywords: Colonoscopy; Colonoscopy preparation; screening; New media; SMS; Short message service
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS receiving (Active Comparator): Study participants of the SMS group receive in total 14 short messages (SMS) containing time adjusted information on colonoscopy preparation starting 4 days before colonoscopy appointment on their mobile phones.
  Interventions: Procedure: Colonoscopy; Device: mobile phone
- Non-SMS receiving (Active Comparator): Study participants of the Non-SMS-Group do not receive any SMS before colonoscopy. Preparation is done according to regular written information given to the patient.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy is performed in both study arm as standard examination
Device: mobile phone — SMS received by mobile phone
  Arms: SMS receiving

SUMMARY:
The purpose of this study is to analyze if integration of new media (SMS) could improve the quality of colonoscopy preparation.

DETAILED DESCRIPTION:
The study approach is the implementation of new media into colonoscopy preparation. As most of our patients already use mobile phones the study should evaluate if time adjusted information about diet recommendation, laxative intake and behavioral recommedation improve the patient compliance and the quality of colonoscopy preparation. In total 14 SMS wil be sent to the study participants starting 4 days prior the colonoscopy appointment. No additional or different information is provided in comparison to regular colonoscopy preparation for out-patient colonoscopy.

Study participant are randomized when included into the study. Group 1 receives a SMS- supported colonoscopy preparation, group 2 receive no SMS and prepares regularly.

Primary endpoint is bowel cleanness measured by Boston Bowel preparation scale, secondary endpoints are patient satisfaction, adenoma detection rate and compliance.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* written informed consent
* mobile phone user
* appointment for outpatient colonoscopy

Exclusion Criteria:

* no outpatient colonoscopy
* no mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-12; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Bowel cleanness measured by Boston Bowel preparation Scale | 1 day
  Boston bowel preparation scale (BBPS) is measured by the endoscopist during colonoscopy

SECONDARY OUTCOMES:
Adenoma detection rate | 1 day
  Histopathological analysis of polyps resected towards adenoma rate
Patient satisfaction and compliance | 1 day
  Patient´s satification with the colonoscopy preparation either SMS supported or not ist asked by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Walter, MD, Principal Investigator — Physician
Locations (4):
- Germany (4):
  - Dr. Aschenbeck, Berlin
  - Gastroenterologische Praxis Prof. Leopold Ludwig, Dornstadt
  - II. Medizinische Klinik Krankenhaus Landshut-Achdorf, Landshut
  - 2nd Medical Department, Klinikum rechts der Isar, Munich

REFERENCES:
- [Derived] Walter B, Klare P, Strehle K, Aschenbeck J, Ludwig L, Dikopoulos N, Mayr M, Neu B, Hann A, Mayer B, Meining A, von Delius S. Improving the quality and acceptance of colonoscopy preparation by reinforced patient education with short message service: results from a randomized, multicenter study (PERICLES-II). Gastrointest Endosc. 2019 Mar;89(3):506-513.e4. doi: 10.1016/j.gie.2018.08.014. Epub 2018 Aug 21. PMID 30138612